CLINICAL TRIAL: NCT06540352
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel Group Study to Select the Dose and Evaluate the Effectiveness and Safety of the Drug Refralon®, Tablets, 1 mg (Pharmproekt JSC) for Long-term Use to Prevent Recurrence of Atrial Fibrillation/Flutter After Terminating Its Persistent Form
Brief Title: A Study to Select the Dose and Evaluate the Effectiveness and Safety of the Drug Refralon®, Tablets, 1 mg for Long-term Use to Prevent Recurrence of Atrial Fibrillation/Flutter After Terminating Its Persistent Form
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Medical Research Center for Cardiology, Ministry of Health of Russian Federation (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: REF-II-08-2023
Record Dates: First submitted 2024-08-01; First posted 2024-08-06 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Atrial Fibrillation; Atrial Flutter
Keywords: Refralon; Cavutilide; Niferidil; class III antiarrhythmic drug; new Russian drug; atrial fibrillation (AF); tablet; atrial flutter (AFL)
MeSH Terms: conditions — Atrial Fibrillation; Atrial Flutter | interventions — Mannitol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator)
  Interventions: Drug: Mannitol
- 1 mg (Experimental)
  Interventions: Drug: 4-Nitro-N-[(1RS)-1-(4-fluorophenyl)-2-(1-ethylpiperidin-4-yl)ethyl]benzamide hydrochloride
- 2 mg (Experimental)
  Interventions: Drug: 4-Nitro-N-[(1RS)-1-(4-fluorophenyl)-2-(1-ethylpiperidin-4-yl)ethyl]benzamide hydrochloride

INTERVENTIONS:
Drug: 4-Nitro-N-[(1RS)-1-(4-fluorophenyl)-2-(1-ethylpiperidin-4-yl)ethyl]benzamide hydrochloride — The drug Refralon® (n-1-[(4-fluorophenyl)-2-(1-ethyl-4-piperidyl)-ethyl]-4-nitrobenzamide hydrochloride) in the dosage form of a concentrate for the preparation of a solution for intravenous administration is registered for medical use in RF June 24, 2014, re-registration was successfully completed on November 20, 2019, registration certificate LP 002510, until December 31, 2025.
  Arms: 1 mg; 2 mg
Drug: Mannitol — Placebo in tablets
  Arms: Placebo

SUMMARY:
Refralon® tablets in two different doses (1 or 2 tablets per day) will be evaluated vs. placebo in patients with persistent atrial fibrillation/flutter after synus rhythm restoration in order to prevent recurrence of arrhythmia. Efficacy and safety of Refralon® tablets will be studied, its optimal dose will be selected and its pharmacokinetics will be evaluated in 14 days, 1, 3 and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Persistent form of AF/AFL lasting 7 days - 1 year (including patients who have previously undergone ineffective catheter or surgical ablation of AF or AFL and patients with a pacemaker or implanted cardioverter-defibrillator (ICD));
* Basic rhythm - AF and/or AFL according to the results of 12-lead ECG at randomization (Visit 2);
* Left ventricular ejection fraction (LVEF) >40% according to the Simpson method;

Exclusion Criteria:

* Intake of class IA, IC and class III antiarrhythmic drugs less than 7 days (for amiodarone less than 60 days) before the study drug intake;
* History of myocardial infarction or other structural heart disease;
* QT prolongation over 500 ms.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-06-03 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects in the group who were shown to maintain sinus rhythm at the end of 6 months of follow-up; | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- National Medical Research Center for Cardiology, Ministry of Health of Russian Federation Organization, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Beliaeva MM, Dzaurova KM, Yuricheva YA, Novikov PS, Mironov NY, Tarasovskiy GS, Zelberg MA, Sokolov SF, Golitsyn SP. Intravenous Cavutilide for Pharmacological Conversion of Paroxysmal and Persistent Atrial Fibrillation in Patients with Heart Failure. J Cardiovasc Dev Dis. 2023 Dec 6;10(12):487. doi: 10.3390/jcdd10120487. PMID 38132655
- [Background] Abramochkin DV, Pustovit OB, Mironov NY, Filatova TS, Nesterova T. Characterization of hERG K+ channel inhibition by the new class III antiarrhythmic drug cavutilide. Naunyn Schmiedebergs Arch Pharmacol. 2024 Jul;397(7):5093-5104. doi: 10.1007/s00210-023-02940-5. Epub 2024 Jan 15. PMID 38224347
- [Background] Egorov YV. Atypical Antiadrenergic Effect of Refralon as a Mechanism of High Antiarrhythmic Effectiveness. Bull Exp Biol Med. 2024 May;177(1):57-62. doi: 10.1007/s10517-024-06131-x. Epub 2024 Jul 2. PMID 38954299
- [Background] Gagloeva DA, Dzaurova KM, Zelberg MA, Mironov NY, Yuricheva YA, Sokolov SF, Golitsyn SP. Early initiation of anti-relapse antiarrhythmic therapy in patients with atrial fibrillation and flutter after pharmacological cardioversion with refralon. Kardiologiia. 2023 Jun 30;63(6):21-27. doi: 10.18087/cardio.2023.6.n2276. English, Russian. PMID 37470730
- [Background] Abramochkin DV, Pustovit OB, Mironov NY, Filatova TS, Kuzmin VS. The Dependence of the Electrophysiological Effects of Class III Antiarrhythmic Drug Refralon on the Frequency of Myocardium Activation. Bull Exp Biol Med. 2023 Mar;174(5):610-615. doi: 10.1007/s10517-023-05756-8. Epub 2023 Apr 11. PMID 37040036
- [Background] Dzaurova KM, Mironov NY, Yuricheva YA, Vlodzyanovsky VV, Mironova NA, Laiovich LY, Malkina TA, Zinchenko LV, Sokolov SF, Golitsyn SP. [Efficiency and safety of using the modified protocol for the administration of the domestic class III antiarrhythmic drug for the relief of paroxysmal atrial fibrillation]. Ter Arkh. 2021 Sep 15;93(9):1052-1057. doi: 10.26442/00403660.2021.09.201008. Russian. PMID 36286864
- [Background] Golitsyn SP, Saidova MA, Sokolov SF, Vlodzyanovskiy VV, Malkina TA, Rozenshtraukh LV, Chazov EI. [Restoration of Sinus Rhythm in Patients With Persistent Atrial Fibrillation and Obesity: New Possibilities of Pharmacological Cardioversion]. Kardiologiia. 2017 Oct;57(10):80-86. doi: 10.18087/cardio.2017.10.10036. Russian. PMID 29276933
- [Background] Maykov EB, Yuricheva YA, Mironov NY, Sokolov SF, Golitsyn SP, Rozenshtraukh LV, Chazov EI. [Refralon (niferidil) is a new class III antiarrhythmic agent for pharmacological cardioversion for persistent atrial fibrillation and atrial flutter]. Ter Arkh. 2015;87(1):38-48. doi: 10.17116/terarkh201587138-48. Russian. PMID 25823268
- See also: Russian registry of clinical trials record — https://grlsbase.ru/clinicaltrails/clintrail/13601